CLINICAL TRIAL: NCT00172549
Title: Quality of Life and Its Related Factors of Patients With Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701176
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study was to explore the quality of life and its related factors of patients with major depressive disorder. This study adopted cross-sectional research design. Purposive sampling was used to collect data from 120 patients came from the psychiatric outpatient departments of a medical center and a psychiatric hospital in northern Taiwan. Data were collected through structured questionnaires, which included：(1) demographic data sheet, (2) 5-item Brief Symptom Rating Scale (BSRS-5), (3) the Center For Epidemiologic Studies Depression Scale(CES-D), (4) Inventory of Socially Supportive Behaviors(ISSB), (5) World Health Organization's Questionnaire on Quality of Life：BREF-Taiwan Version 100(WHOQOL-BREF). Data were analyzed by using SPSS/Windows 10.0 statistical software. The descriptive statistics methods included frequency distribution, arithmetic mean, standard deviation, and percentage. Data were analyzed by using independent t-test, Pearson's product-moment correlation, one way ANOVA and stepwise multiple regression and so on, with which we can examine the demographic, degree of depression, social support and their links to the quality of life. Through the research, we found out the following results：

1.The condition of major depressive disorder patients' quality of life is score range of each subtitle from 4-20. A sum from the following subtitles：physical domain is 11.54, psychological domain is 10.46, social domain is 11.61 and environmental domain is 12.82. The quality of life results is higher of environmental domain, which is poorer of psychological domain.

2. The results of quality of life related to demographic, degree of depression, social support were as followed：

1. Physical domain：the independent variables of significant linear correlation is age, the age of early-onset, type of occupation, living arrangements, economic status, health status, the degree of depression and emotional support.
2. Psychological domain：the independent variables of significant linear correlation is age, the age of early-onset, type of occupation, living arrangements, economic status, health status, the degree of depression, the sum of social support, emotional support, instrumental support, informational and appraisal support.
3. Social domain：the independent variables of significant linear correlation is age, the age of early-onset, marital status, type of occupation, economic status, health status, the degree of depression, the sum of social support, emotional support, instrumental support, informational and appraisal support.
4. Environmental domain：the independent variables of significant linear correlation is age, the age of early-onset, marital status, economic status, the degree of depression, the sum of social support and emotional support.

3.The best stepwise regression models of predicting major depressive disorder patients' quality of life were as followed：

1. Physical domain：the best predicting factor is the degree of depression, and accounted for explained 60.30﹪of the variance.
2. Psychological domain：the best predicting factors are the degree of depression, the sum of social support, the age of early-onset, age more than 71 years old, and accounted for explained 76.50﹪of the variance.
3. Social domain：the best predicting factors are the degree of depression, the age of early-onset, informational and appraisal support, unemployment and age more than 71 years old, and accounted for explained 53.80﹪of the variance.
4. Environmental domain：the best predicting factors are the degree of depression, income less than one hundred thousand, income more than one hundred ten thousand and more than 71 years old, and accounted for explained 53.50﹪of the variance.

The results of this study could understand major depressive disorder patients' quality of life condition and provide related research in the future, develop local data and health administration reference of foundation.

ELIGIBILITY:
Inclusion Criteria:

* people with Major Depressive Disorder

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2004-03; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Chuan Hsiung, Ph.D, Study Chair — Department of Nursing, National Taiwan University